CLINICAL TRIAL: NCT02228733
Title: An Open-Label, Parallel-Group, Single Ascending Dose Study in Healthy Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of KBP-5074 Following Oral Administration and With a Food Effect Panel
Brief Title: Phase 1 Single Ascending Dose Study to Evaluate Safety, Tolerability and Pharmacokinetics of KBP-5074
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBP5074-1-001
Record Dates: First submitted 2014-08-25; First posted 2014-08-29 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — KBP-5074

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- KBP-5074: Cohort 1 (Experimental): Healthy Volunteers will receive one dose of KBP-5074
  Interventions: Drug: KBP-5074
- KBP-5074: Cohort 2 (Experimental): Healthy Volunteers will receive one dose of KBP-5074
  Interventions: Drug: KBP-5074
- KBP-5074: Cohort 3 (Experimental): Healthy Volunteers will receive one dose of KBP-5074
  Interventions: Drug: KBP-5074
- KBP-5074: Cohort 4 (Experimental): Healthy Volunteers will receive one dose of KBP-5074
  Interventions: Drug: KBP-5074
- KBP-5074: Cohort 5 (Experimental): Healthy Volunteers will receive one dose of KBP-5074
  Interventions: Drug: KBP-5074
- KBP-5074: Fed Group (Experimental): Healthy Volunteers will receive one dose of KBP-5074
  Interventions: Drug: KBP-5074

INTERVENTIONS:
Drug: KBP-5074 — Comparisons of different doses of study drug

SUMMARY:
This single ascending dose (SAD) study in healthy subjects will evaluate the safety, tolerability and pharmacokinetics of KBP-5074. PK/PD (plasma aldosterone, serum potassium and urine albumin levels) relationships will be explored to support the selection of dosing regimens of KBP-5074 that are suitable for the Phase 2 dose-finding study to evaluate the efficacy, safety and tolerability of KBP-5074 in patients that could slow the progression of nephropathy as well as control hypertension.

DETAILED DESCRIPTION:
This is an open-label, parallel-group, dose-escalation study to evaluate the safety, tolerability and pharmacokinetics of KBP-5074 following a single dose administration of KBP-5074 with and without food. The study includes 2 parts.

Part 1: Pharmacokinetics from each dose cohort will be characterized before initiation of dosing in the subsequent cohorts. Eight subjects in each dose cohort will receive active drug. The total number of cohorts will be up to 5. Extensive PK samplings will be collected prior to and following administration of single dose of KBP-5074.

Part 2: A separate panel of 6 subjects will receive a single dose of KBP-5074 under fed conditions. Extensive PK samplings will be collected prior to and following administration of single dose of KBP-5074 under fed conditions.

Serum and plasma samples for pharmacodynamic markers (plasma aldosterone and serum potassium levels) will be collected at pre-dose and postdose in both Part 1 and Part 2.

The urine samples will be also used for quantitative determination of urinary albumin in both Part 1 and Part 2.

Safety assessments will include monitoring of adverse events (AEs), vital signs (blood pressure, pulse rate, respiratory rate and oral temperature), clinical laboratory findings, 12-lead electrocardiograms (ECGs), and physical examination findings.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 19 ≤ BMI ≤ 30 kg/m2, no significant medical history, normal renal function and in good general health

Exclusion Criteria:

* Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity; A history of prescription drug abuse, or illicit drug use within 6 months prior to screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability | 14 days
  Assessing the number of participants with adverse events, abnormal vital signs, clinical laboratory findings, 12-lead ECGs and physical examinations): pre dose and post dose
Area Under Curve (AUC) Time Frame | 14 days
  Assessing drug exposure across time. AUC is a useful metric when trying to determine whether two formulations of the same dose (for example a capsule and a tablet) result in equal amounts of tissue or plasma exposure. Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120, 168, 216, 264 and 312 hours post-dose

SECONDARY OUTCOMES:
The effect of food on Area Under Curve (AUC) Time Frame | 14 days
  Assessing the food effect on drug exposure across time at pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120, 168, 216, 264 and 312 hours post-dose
The plasma aldosterone, serum potassium and urine albumin levels | 14 days
  Assessing blood levels of aldosterone, potassium and urine albumin at pre dose and postdose